CLINICAL TRIAL: NCT02095717
Title: Multicenter Study Comparing Taxotere Plus Curcumin Versus Taxotere Plus Placebo Combination in First-line Treatment of Prostate Cancer Metastatic Castration Resistant (CURTAXEL)
Acronym: CURTAXEL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was stopped for futility in view of the results of the interim analysis
Sponsor: Centre Jean Perrin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013-002138-20
Record Dates: First submitted 2014-03-20; First posted 2014-03-26 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Prostate Cancer Metastatic Castration Resistant
MeSH Terms: interventions — Curcumin; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Curcumin (Experimental): curcumine capsule
  Interventions: Drug: Curcumin; Drug: Taxotere
- Placebo (Placebo Comparator): placebo capsule
  Interventions: Drug: Placebo; Drug: Taxotere

INTERVENTIONS:
Drug: Curcumin
  Arms: Curcumin
Drug: Placebo
  Arms: Placebo
Drug: Taxotere

SUMMARY:
Multicenter randomized phase II study, double-blind, comparing Taxotere plus curcumin versus Taxotere plus placebo combination in first-line treatment of prostate cancer metastatic castration resistant. Assess time to progression (time to progression) of metastatic disease (from first day of treatment in the trial).

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years.
* Performance status ≤ 2 according to the WHO criteria.
* Life expectancy> 3 months.
* Patient in hormonal blockade based on surgical castration by orchiectomy or pulpectomy, medical or agonist or antagonists of LHRH associated or not with anti-androgens or any other treatment that blocks the fraction of non-gonadal testosterone, resulting in a testosterone <0.5 ng / mL.
* Patient with adenocarcinoma of the prostate and histologically proven metastatic castration-resistant stage, defined by: objective progression of at least one measurable tumor target and / or assessable by RECIST, and / or increase in PSA ("rising PSA").
* Satisfactory biological functions (renal, hepatic and hematologic)
* Patient who signed the consent for participation before entering the study.
* Affiliation to a social security scheme (or be the beneficiary of such a plan) under the terms of the law of 9 August 2004.

Exclusion Criteria:

* Age <18 years.
* Performance status> 2 according to the WHO criteria.
* Patient deprived of liberty or under guardianship, patient with (the) condition (s) psychological, family, social or geographic may interfere with the proper conduct of the study.
* Diagnosis of a second malignancy in the past 5 years, with the exception of a basal cell skin cancer considered cured.
* Patient with brain metastases at initial assessment.
* Patient with another pathology deemed incompatible with the inclusion in the protocol.
* Laboratory tests inadequate.
* History of malabsorption syndrome or extensive resection of the upper digestive tract.
* Uncontrolled intercurrent infection.
* Pathology autoimmune and / or chronic active inflammation.
* peripheral neuropathy grade 2 according to the criteria of the National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE, version 4.0).
* History of allergy to polysorbate 80.
* Treatment with nonsteroidal anti-inflammatory and / or cyclooxygenase-2 dated within three weeks.
* Concomitant with a drug test or participation in another clinical trial within <30 days treatment.
* Regular Taking dietary supplements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Time to progression | participants will be followed post treatment. From date of randomization until the date of first documented progression or date of death from any cause
  Assess time to progression (time to progression) of metastatic disease (from first day of treatment in the trial). Progression was defined as an increase (of) injury (s) tumor (s) (RECIST) or an increase in PSA levels (≥ 25% and ≥ 2ng/ml increase) or the appearance of new lesions metastatic (at least 2 new lesions for bone lesions).
  From date of randomization until the date of first documented progression or date of death from any cause

SECONDARY OUTCOMES:
PSA response | From date of randomization until the date of first documented PSA progression or date of death from any cause
  Evaluate the PSA response (50% decrease compared to the initial value)
objective tumor response rate | participants will be evaluated at the end of the treatment (randomization + an expected average of 4 months)
  Evaluate the objective tumor response rate (CR + PR) by RECIST.
safety and tolerability | patients will be followed for the duration of the treatment, an expected average of 4 months
  Assess the safety (adverse events) of the combination Taxotere/ curcumin.
Pain | participants will be followed at Cycle1,3,6 of chemotherapy and post treatment (+1months after the end of the treatment)
  Assess pain in the short questionnaire on pain (QCD)
neuroendocrine markers | participants will be followed for the duration of the treatment, an expected average of 4 months
  Assess serum neuroendocrine markers
Overall survival | from date of randomization until the date of death from any cause
  Evaluate overall survival (between inclusion and death whatever the cause)
anti-angiogenic activity | participants will be followed at each Cycle of chemotherapy ( + inclusion) , an expected average of 4 months
  Evaluate the anti-angiogenic activity of the association Taxotere ® plus curcumin
compliance | patients will be followed for the duration of the treatment, an expected average of 4 months
  Assess the compliance by curcumin treatment / placebo orally

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Clinique de la Chataigneraie, Beaumont
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay
  - Institut Jean Godinot, Reims